CLINICAL TRIAL: NCT03532529
Title: Evaluation of Speckle Tracking Parameters as Predictors of Successful VA ECMO Weaning Procedure. A Prospective Observational Pilot Study.
Brief Title: Evaluation of Speckle Tracking Parameters as Predictors of Successful VA SPECKLE ECMO
Acronym: SPECKLE-ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 241001
Record Dates: First submitted 2018-05-10; First posted 2018-05-22 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experiencing the composit outcome: Average values of LV longitudinal strain^ (Midesophageal 4 chamber view) in patients who developed the composite outcome including the following outcomes of interest:
  * death within 30 days from VA ECMO liberation
  * the necessity of new Mechanical Circulatory Support (VA-ECMO, Impella, LVAD) within 30 days from VA ECMO liberation
    o Whether after VA ECMO liberation the patient still needs IABP or a RVAD support, this situation is not considered necessity of new Mechanical Circulatory Support. A necessity of new Mechanical Circulatory Support is defined when IABP or RVAD or VA ECMO or Impella are needed again after their removal
  * heart transplantation within 30 days from VA ECMO liberation
  Interventions: Other: not applicable, it is an observational study
- not experiencing the composit outcome: Average values of LV longitudinal strain^ (Midesophageal 4 chamber view) in patients who did not develop the composite outcome including the following outcomes of interest:
  * death within 30 days from VA ECMO liberation
  * the necessity of new Mechanical Circulatory Support (VA-ECMO, Impella, LVAD) within 30 days from VA ECMO liberation
    o Whether after VA ECMO liberation the patient still needs IABP or a RVAD support, this situation is not considered necessity of new Mechanical Circulatory Support. A necessity of new Mechanical Circulatory Support is defined when IABP or RVAD or VA ECMO or Impella are needed again after their removal
  * heart transplantation within 30 days from VA ECMO liberation
  Interventions: Other: not applicable, it is an observational study

INTERVENTIONS:
Other: not applicable, it is an observational study — not applicable, it is an observational study

SUMMARY:
Purpose of this study is to assess whether measurements obtained through speckle tracking (LV longitudinal and circumferential strain, RV longitudinal strain) can give additional information in identifying patients who develop adverse outcomes 30 days post successfully weaning from VA ECMO (liberation not for palliation). It is a prospective observational non-blinded pilot study.

In order to achieve this purpose, speckle tracking analysis will be performed on the recorded images of the transoesophageal echocardiogram performed during the last VA ECMO weaning study of patients defined ready for VA ECMO liberation. VA ECMO liberation will be based according to LVOT VTI increase and clinical judgment during patients' VA ECMO weaning study. It will be assessed whether the population experiencing the outcomes of interest (death within 30 days from VA ECMO liberation, hospital admission for a new episode of cardiogenic shock or heart failure within 30 days from VA ECMO liberation, need for new mechanical circulatory support within 30 days from VA ECMO liberation) and the population not experiencing these outcomes have different values of strain (LV longitudinal and circumferential and RV longitudinal strain) during the weaning study.

DETAILED DESCRIPTION:
This project is non-commercial study which aims to assess whether measurements derived through speckle tracking give additional information to conventional echocardiographic parameters (LVOT VTI measurements, etc.) in identifying patients at greatest risk of major clinical events occurring within 30 days after VA ECMO liberation. It is a prospective observational non-blinded pilot study. In this study will be investigated whether particular values of strain (longitudinal and circumferential LV longitudinal and circumferential and RV longitudinal strain) and conventional echocardiographic parameters, obtained during VA ECMO weaning studies, are more associated to major clinical outcomes within 30 days after VA ECMO liberation.

The population consists of patients receiving VA ECMO mechanical circulatory support for cardiogenic shock, who have undergone an echocardiogram as part of the weaning process and a decision has been made to attempt weaning from VA ECMO. The decision to wean the patient from VA ECMO will be made by the attending clinician who will be aware of all echocardiographic measurements with the exception of the speckle tracking results (as is the standard-of-care at our institution). The study investigator who will perform all speckle tracking analysis will not be involved in the decision to wean from VA ECMO.

SCHEMATIC OF STUDY DESIGN

1. Screening of VA ECMO patients in whom a weaning study is planned
2. Definitive SCREENING FAILURE = patients who do not fulfil inclusion criteria or have at least one exclusion criterion (not including the LVOT VTI criterion)
3. VA ECMO weaning study performed

   * Patients deemed unsuitable for liberation from VA ECMO at this time are not enrolled for analysis, and are reassessed following the next weaning study
   * Patients deemed suitable for liberation from VA ECMO, but whose LVOT VTI was <10cm at any stage of the weaning study, or whose LVOT VTI at lowest achieved flow was lower than baseline are excluded
   * Patients deemed suitable for liberation from VA ECMO and not excluded based on LVOT VTI criterion are enrolled.
4. EVALUATION OF SPECKLE TRACKING FINDINGS (LV LONGITUDINAL AND CIRCUMFERENTIAL AND RV LONGITUDINAL STRAIN) AND CONVENTIONAL ECHOCARDIOGRAPHIC PARAMETERS WITH CLINICAL OUTCOMES AT 30 DAYS POST VA ECMO LIBERATION (REMOVAL)

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years.
* Receiving VA ECMO mechanical circulatory support for cardiogenic shock and planning to undergo an echocardiogram as part of a VA ECMO weaning study.
* Informed consent for study participation provided by the patient (where able) or personal consultee (where the patient is unable to provide consent) or nominated consultee (where the patient is unable to provide consent and no personal consultee is available).

Exclusion Criteria:

* Contraindication to transoesophageal echocardiography.
* Patients who are expected to require heart transplantation, LVAD or biventricular VAD within 30 days from admission.
* Patients who are not expected to survive weaning from VA ECMO (liberation from VA ECMO exclusively for purpose of palliation).
* Contemporary presence of Impella device during VA ECMO weaning study.
* Patients in atrial fibrillation or in a different rhythm from sinus at the moment of VA ECMO weaning study.
* Patient's LVOT VTI is less than 10cm at any stage of VA ECMO weaning study and/or LVOT VTI is lower at the lowest achieved blood flow than it was at baseline (LVOT VTI criterion).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients admitted to the ICU requiring mechanical circulatory support with VA ECMO and a diagnosis of cardiogenic shock (of any aetiology) who recover cardiac function to the point of decision to liberate (to wean) from VA ECMO.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-11-28 (Estimated); Study Completion 2019-11-28 (Estimated)

PRIMARY OUTCOMES:
the composite outcome | within 30 days from VA ECMO liberation
  the composite outcome including the following outcomes of interest:
  * death within 30 days from VA ECMO liberation
  * the necessity of new Mechanical Circulatory Support (VA-ECMO, Impella, LVAD) within 30 days from VA ECMO liberation
    o Whether after VA ECMO liberation the patient still needs IABP or a RVAD support, this situation is not considered necessity of new Mechanical Circulatory Support. A necessity of new Mechanical Circulatory Support is defined when IABP or RVAD or VA ECMO or Impella are needed again after their removal
  * heart transplantation within 30 days from VA ECMO liberation

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital and Harefield NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided